CLINICAL TRIAL: NCT06788028
Title: Optimizing Multi-level Interventions to Improve Child Mental Health in Azerbaijan
Brief Title: Multi-level Child Mental Health Interventions in Azerbaijan
Acronym: AZ CMH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IRB24-1074; R01MH135095 (NIH)
Record Dates: First submitted 2024-12-31; First posted 2025-01-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Mental Health; Child Externalizing Problems; Child Behavior Problem
Keywords: Azerbaijan; Children; Child Mental Health; Family Strengthening; Economic Empowerment; Child and Family Well-being
MeSH Terms: conditions — Psychological Well-Being | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: The study will use a randomized design and apply MOST approach to test and compare the three intervention components: a) a family-strengthening intervention (yes or no); b) trauma-focused mental health services (yes or no); and c) economic empowerment in the form of Child Savings Accounts /Child Development Accounts-CDAs (yes or no). There are three factors (intervention components) and each factor has two levels. This is a 2*2*2, or 23, factorial design and, therefore, the study will have eight different experimental conditions or groups (2*3 = 8). All participating families are eligible to receive the government-based usual care.
  The eligible and consenting child-parent dyads (N=600) will be randomly assigned to one of eight study groups, determining how many and which intervention components participants will receive. Given this design, half of the sample will receive each intervention component.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Family Strengthening, Mental Health, Economic Empowerment (Experimental): Group will receive: 1) Usual Care, 2) Family Strengthening, 3) Trauma-focused Mental Health Services, and 4) Economic Empowerment Interventions
  Interventions: Behavioral: Family Strengthening; Behavioral: Mental Health Screening, Referral and Connection to Services; Other: Economic Empowerment
- Family Strengthening, Mental Health (Experimental): Group will receive: 1) Usual Care, 2) Family Strengthening, and 3) Trauma-focused Mental Health Services
  Interventions: Behavioral: Family Strengthening; Behavioral: Mental Health Screening, Referral and Connection to Services
- Family Strengthening, Economic Empowerment (Experimental): Group will receive: 1) Usual Care, 2) Family Strengthening, and 3) Economic Empowerment Interventions
  Interventions: Behavioral: Family Strengthening; Other: Economic Empowerment
- Family Strengthening Only (Experimental): Group will receive: 1) Usual Care and 2) Family Strengthening Interventions
  Interventions: Behavioral: Family Strengthening
- Mental Health, Economic Empowerment (Experimental): Group will receive: 1) Usual Care, 2) Trauma-focused Mental Health Services, and 3) Economic Empowerment Interventions
  Interventions: Behavioral: Mental Health Screening, Referral and Connection to Services; Other: Economic Empowerment
- Mental Health Only (Experimental): Group will receive: 1) Usual Care and 2) Trauma-focused Mental Health Services
  Interventions: Behavioral: Mental Health Screening, Referral and Connection to Services
- Economic Empowerment Only (Experimental): Group will receive: 1) Usual Care and 2) Economic Empowerment Interventions
  Interventions: Other: Economic Empowerment
- Usual Care Only (Experimental): Group will receive: Usual Care Intervention only
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Usual Care — All participants receive the usual care via standard mental health services offered by the NMHC to the public free of charge. Participants will have access to these public services regardless of whether or not they choose to participate in this study. If they refuse to participate in the research study, they will still have access to usual care.
  Arms: Usual Care Only
Behavioral: Family Strengthening — Families will engage in 12 weekly (1-1.5 hours) of family strengthening sessions, led by trained facilitators from the Research and Education Center. Groups will be composed of approximately 5 caregiver-child dyads. Sessions are designed to improve family functioning, strengthen child-parent relationships, enhance parenting strategies, and prevent emotional and behavioral problems among at-risk children.
  Arms: Family Strengthening Only; Family Strengthening, Economic Empowerment; Family Strengthening, Mental Health; Family Strengthening, Mental Health, Economic Empowerment
Behavioral: Mental Health Screening, Referral and Connection to Services — Children will receive 12 sessions of individual mental health services. Clinicians are trained in the Attachment, Regulation, and Competency (ARC) framework. Services include a clinical assessment performed by a psychiatrist, development of an individual care plan, and corresponding mental health services, informed by ARC.
  Arms: Family Strengthening, Mental Health; Family Strengthening, Mental Health, Economic Empowerment; Mental Health Only; Mental Health, Economic Empowerment
Other: Economic Empowerment — Child Development Accounts (CDAs) will be opened to facilitate family savings. The project will provide $50 as seed money to open a savings account in the child's name. Savings of up to $20 per month will be matched with study funds at a rate of 2:1 and placed in the CDA account. Caregivers and children will also engage in 12 weekly (1-1.5 hours) of financial education sessions, led by facilitators from the Research and Education Center.
  Arms: Economic Empowerment Only; Family Strengthening, Economic Empowerment; Family Strengthening, Mental Health, Economic Empowerment; Mental Health, Economic Empowerment

SUMMARY:
To improve mental health outcomes among children aged 7-14 from low-income families in Azerbaijan, this study will refine and test three evidence-based intervention approaches: family-strengthening intervention; trauma-focused mental health services; and economic empowerment in the form of Child Savings Accounts.

Based on prior research on the mental health of deinstitutionalized children conducted by this U.S.-Azerbaijani team in collaboration with a local Community Collaborative Board, these intervention components have been adapted to maximize fit to the cultural context of Azerbaijan. In this study, the adapted interventions will be tested with 600 child-caregiver dyads in a trial using the Multiphase Optimization Strategy (MOST) to compare different intervention components and identify the most optimal combination. Given the limited human and financial resources in low- and middle-income countries (LMICs), it will be important to identify whether each of these interventions is necessary and/or sufficient for improving the mental health of children.

The study will test the effects of each intervention component on children's mental health outcomes (symptoms of depression, anxiety; disruptive behaviors; post-traumatic symptoms;), on associated cognitive and social processes (e.g., attention, emotion recognition bias) and functional outcomes (e.g., academic performance). The study will also examine the mediating pathway associated with each intervention component.

DETAILED DESCRIPTION:
Despite progress in mental health care reforms across Azerbaijan and other post-Soviet countries toward reducing reliance on a medicalized model, the demand for mental health services still far exceeds available resources. Mental health care is largely centered on a pathology-oriented approach, focused on the short-term alleviation of symptoms, and neglectful of the social and environmental drivers of psychological distress. The chronic hardship and economic deprivation many in Azerbaijan face-along with prolonged exposure to multiple traumatic events and adverse childhood experiences following a series of wars, political upheavals, and refugee crises-can severely undermine families' ability to care for their children's emotional and behavioral wellbeing.

To reduce the service gap, there is a critical need to develop a package of comprehensive community-based psychosocial strategies that improve child mental health outcomes associated with poverty and adversity. According to the National Institute of Mental Health/NIMH's Grand Challenges in Global Mental Health, the advancement of prevention and early intervention (Goal B) is a key priority. This study will contribute to the development of innovative interventions and critical knowledge to address these priorities.

The specific aims of the research study are:

Aim 1: To refine, test, and compare the effects of three interventions (family-strengthening; economic empowerment, and trauma-focused mental health care) on mental health clinical outcomes (including internalizing problems--depression, anxiety, post-traumatic symptoms-and externalizing problems-aggressive or disruptive behavior), b) cognitive and social processes associated with these outcomes (e.g., attention, inhibitory control, working memory, emotion recognition bias), and c) functional outcomes (e.g., academic performance, peer relations) among 7-14-year-old children with or at risk of mental health problems in Azerbaijan.

Aim 2: To examine the role of hypothesized intervention mediators (emotion regulation, supportive parenting, stress reactivity, and economic wellbeing) and moderators (age, gender, family structure, combination of intervention components, and symptom severity) in improving child mental health outcomes.

Aim 3: To explore facilitating factors and barriers to implementation and participation in each intervention component (at individual, family, and organizational levels) using qualitative interviews with intervention participants and service providers.

Study procedures:

Participants (600 child-caregiver dyads) will be recruited in three cities in Azerbaijan (Baku, Sumgayit, and Ganja) and will be invited to participate in the study. Participants will be assigned at enrollment to receive only usual care (control) or one or more of the three intervention components (family strengthening, mental health, or economic interventions). Participants will engage in 12 weekly sessions for each intervention. Participants will be asked to complete baseline, 1-year and 2-year follow-up surveys. Additionally, post-intervention qualitative interviews (n=60) conducted after completion of the intervention sessions and follow-up visits will solicit participants' and services providers' experiences with each intervention component.

Participants assigned to receive intervention(s) will receive one or a combination of the following:

1. Family Strengthening: Families will receive 12 weekly sessions led by trained facilitators from the Research and Education Center. Due to its focus on family-strengthening, the study uses the evidence-based intervention 'SAFE Children', which employs a multiple family group format and is designed to improve family functioning, strengthen child-parent relationships and communication, enhance supportive parenting strategies, and prevent emotional and behavioral problems among at-risk children.

   Families assigned to this intervention will receive 12 weekly sessions led by trained facilitators from Research and Education Center, focusing on improving family relations with techniques for communication, problem-solving, managing child's behavior, and maintaining support (e.g., Setting a Fun and Positive Atmosphere, Why Play is Important, Making Family Goals Identifying Family Strengths and Problems, Communication with Children, Communication with Adults, Discipline, Anger and Self-Control, Conflict Resolution, Helping Children with Social Relationships, Family Support-Identifying the Need/Where to Go). The intervention developer Dr. Gorman-Smith (Co-I), will oversee the training and implementation process to ensure fidelity to its core components. The adapted intervention incorporates sessions that address issues faced by families (e.g., stigmatized status in the community). Each session lasts about 1-1.5 hours and will be delivered by facilitator and co-facilitator at the NMHC. Sessions will be offered in the afternoons and/or on weekends to accommodate school and parents' schedules.
2. Economic Empowerment: Families assigned to this intervention will participate in: a) the opening of a matched savings account, b) 12-session financial education for families and c) monthly mentoring sessions.

   1. Child Savings Account: This component will a) connect families to a bank, and b) train families how to save small amounts which will be matched using project funds. The project will provide 85 AZ manat (50 USD) as seed money to open a savings account in each child's name, managed in-trust by a parent or legal guardian. The child's caregiver will make small monthly contributions to this savings account and present bank statements for proof of savings. A savings account for matched savings (Child Development Account-CDA) will be created in each child's name and managed by the Research and Education Center. Savings of up to 34 AZ manat (20 USD) per month in a personal account will be matched with project funds at a 2:1 rate into the matched savings account. For example, if a family deposits 15 AZ manat in their savings account, the study will deposit 30 AZ manat in the matched savings account, as this is a 2:1 match on the original 15 AZ manat deposit. If a family deposits 20 AZ manat in their personal savings account, the study will deposit 40 AZ manat in the matched savings account.

      Matched savings can only be used for "authorized expenses", or expenses towards a child's education (e.g., to pay directly for school expenses), housing (e.g., to rent an apartment), or to start or expand a small family business (e.g., opening a kiosk or beauty/barbershop). Thus, if a family saves 30 AZ manat each month for 12 months, the child will have a total of 1165 AZ manat saved by the end of the pilot study (360 manat in family contributions and 720 manat in matched funds from the project, plus the seed amount of 85 manat). In Azerbaijan, 1100 manat can cover one year of college, an amount generally unattainable for poor families with multiple children.

      If a family wants to use matched funds for an authorized expense, they will submit a withdrawal request to the Research and Education Center. The study coordinator at the Research and Education Center will notify the family if the request has been approved. Families will provide receipts for authorized expenses to be reimbursed by the study via voucher, check or direct transfer to a personal bank account. The matched savings accounts will be managed by the Research and Education Center and matched savings will be added to this account based on the physical monthly bank statements that families share with the study team.

      The personal savings account that was opened at the beginning of the study is managed by the youth's legal guardian (parent) and only a legal guardian may request matched funds for authorized expenses. The study does not have access to this bank account and the only information given to the study team about this account is shared through monthly bank statements that families will bring to the mentoring session and share with their mentor. If families do not bring their bank statements with them to mentoring sessions, the mentor will still discuss financial decision-making, saving and other topics (such as meeting financial goals) with the youth and their caregiver. The mentor will not guide the family on how much to save or withdraw from their account. They will help the family to make decisions to meet the family's financial goals, as determined by the youth and caregiver.

      Matched funds are available to families up to one year after the conclusion of the study the course of the study. Participants will be continually encouraged to use the funds during the study period for several reasons. First, the study team aims to guarantee that matched funds go to allowable expenses that will benefit youth and families. Second, post-intervention follow-up interviews will be conducted and the study team hopes to assess the impact of the intervention, ideally after families have spent the matched funds on allowable expenses. Third, this economic intervention is following the protocol of previous Child Development Account intervention studies which also encourage the use of funds during the study period.
   2. Financial Education Curriculum: Children and their caregivers will participate in training on Savings and Financial Planning. Parents and children will attend separate sessions for 12 weeks, each for one hour. Sessions will be delivered in a group format and led by economic intervention facilitators from the Research and Education Center.

      The parent curriculum will cover: The Importance of Saving; Identifying and Managing Resources; Setting Up a Savings System; Sources of Income; and Budgeting and Spending, Planning for Unexpected. This manual was originally developed by Dr. Ssewamala for Uganda, and has been redesigned, adapted, and tested with low-income families in Azerbaijan. The Research and Education Center (REC) facilitators have received training and guidance on the delivery and monitoring of the intervention. The manual on financial education and entrepreneurship for school children has been translated and adapted jointly with the Junior Achievement-Azerbaijan and tested in the previous study. Dr. Ssewamala, Co-I, will provide additional training and guidance to the REC staff involved in the delivery and monitoring of economic intervention.

      Since this study will test the efficacy of each intervention component separately and not as a bundle, at this stage the savings and financial planning training will be offered separately, not integrated with family strengthening sessions, because due to the nature of MOST trials, some families will receive only one of these intervention components, and others will receive both components.
   3. Mentoring: After completing the curriculum and opening a CDA account, each family will also participate in monthly mentoring sessions provided by economic facilitators, to provide support, guidance and discuss any difficulties each family may be facing in achieving their individual financial and saving plan. Through the mentoring sessions, children and their caregivers will be provided guidance and information on how to use what they have learned during the financial education sessions to maintain their bank account, building their relationship to the banking institution, and continue to accumulate assets beyond the scope of the study. The facilitators of the financial education sessions will also serve as mentors for the mentoring component of the economic empowerment intervention.

   Mentors will be responsible for managing conversations between caregivers and children about using bank accounts and managing finances. Mentors will be prepared to handle difficult conversations about money, as this can be a sensitive topic for families. Throughout the study, mentors will be available to support families as they navigate discussions about money and relationships. Families will share their personal account deposit statements with the study team during mentoring sessions and, based on that amount, funds will be added to the matched savings accounts at a rate of 2:1 up to 34 AZ manat (20 USD). Mentors will use a mentoring session planning tool to guide the mentoring sessions and support the family as they save and manage their financial goals. This tool will not be used as a data collection tool. In the case that mentors/facilitators choose to end their participation in the study, other consenting mentors/facilitators will work with parent-child dyads. Mentors will also be responsible for reminding participants of the deadline to spend their matched funds, and offer notices to spend the funds before the time-frame ends.
3. Trauma-focused Mental Health Services: Families assigned to this intervention will receive trauma-focused mental health care informed by the Attachment, Regulation, and Competency (ARC) framework. Services include a clinical assessment performed by a psychiatrist, development of an individual care plan, and connection to the assigned clinician (e.g., a child psychologist, child psychiatrist, or other mental health specialists) to receive corresponding mental health services, informed by ARC. ARC is a flexible, core components framework focused on psycho-education, caregiver affect management, and routines to effectively manage emotional and physiological experiences. This will include 12-individual sessions provided by clinicians at the National Mental Health Center (NMHC), who have received training and use this modality in a previous R01. The NMHC clinicians delivering the intervention will not be involved in the research activities. The research team (e.g., research assistants, project coordinator) will be responsible for referring study participants who have been randomized to this condition to mental health services. If upon review by a leading clinician, the treatment goals have not been achieved, the services can be extended.

Randomization:

Eligible and consenting child-caregiver dyads will be randomized into one of eight experimental conditions. Random digits will be drawn by the PI to assign to order the 8 experimental conditions within each city. Given that two interventions (family strengthening and economic) are group-based, the randomization will be performed in cohorts consisting of 5 families. After the first five families are recruited, the cohort is closed and this group will receive the first ordered experimental condition (e.g., Group #7 economic intervention alone). To minimize any coercion to join the study just for financial reasons, eligible and consenting participants will be informed about the randomized intervention condition upon completion of the baseline interview.

The control group (no intervention) will have access to participate in any of the programs (excluding opening a Child Development Account (CDA) two years after the start of the study.

Assessment:

Youth and caregivers will participate in baseline, 1-year, and 2-year follow-up surveys to assess outcomes and mediator variables. Electronic surveys via Qualtrics will be administered by research assistants to both youth and caregivers and will take about 50 minutes. At the end of each intervention session, participants will also complete a process measure survey including information on participant feedback, satisfaction and perceived usefulness. Assessments will ask about child outcomes (social-emotional, behavioral), mediators (caregiver-child relationships, parental distress, parenting stress, economic wellbeing) and moderators (adverse childhood experiences, socio-demographic characteristics).

Finally, participants will complete follow-up post-intervention qualitative interviews 12 months after the start of the research study. The questions for this interview have not yet been developed. Interview guides will be developed based on the results of the first phase of the study. The PI will submit an amendment to the IRB protocol prior to the beginning qualitative interviews, outlining procedures, consent and administration procedures.

ELIGIBILITY:
Inclusion Criteria:

1. The child is between ages 7 and 14;
2. The child is at-risk for mental health problems as measured by one of the following criteria:

   1. Elevated child emotional behavioral problems as indexed by 'high' or 'very high' scores on the Strengths and Difficulties Questionnaire (SDQ, total difficulty score or any of the four difficulty subscales - emotional, conduct, hyperactivity, or peer problems); OR
   2. Parental risk factor - parental elevated emotional distress, as indexed by 'severe' or 'extremely severe" score on any of the DASS-21 subscales (DASS-21 Stress = 27; Anxiety = 15; or Depression = 15);
3. The child and parent (or other primary caregiver) can commit to study participation.

If a family has more than one eligible child, participation in the study will be offered to the older child. If both the eligible child and caregiver provide consent, they will be enrolled in the study.

All eligible children within a family can be enrolled in the study.

Exclusion Criteria:

Participants will be excluded from participation in the study if the child, the parent or the participating caregiver is assessed to have a cognitive impairment that would interfere with their ability to provide informed consent. This will be assessed during the consent process. As part of the informed consent process, conducted through an Azeri speaking research assistant, potential participants will also be asked to state their understanding of areas addressed during the informed consent discussion including (1) the nature and extent of participation in the study; (2) risks involved with participation; and (3) the potential benefits of participation in the study. If a participant is unable to respond to any of the three items, this youth/caregiver pair will be excluded from the study.

Children and parents will also be excluded if one of them has significant behavioral, and/or mental health impairment (e.g., development disorder, autism, psychosis, high symptoms of trauma or depression) that could interfere with either with their ability to benefit from the prevention program or to participate safely. Research Assistants will ask parents about any of these conditions during the screening process.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in child mental health using the Strengths and Difficulties Questionnaire (SDQ) | Baseline, 12 months, 24 months
  Questions assess child's internalizing problems (depression, anxiety) and externalizing problems (aggressive or disruptive behavior). Strengths and Difficulties Questionnaire includes five scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behaviors reported by parent/caregiver and teacher. With the exception of prosocial behaviors, a higher score indicates a worse outcome. For the prosocial scale, a higher score indicates a better outcome. The total score minimum value is 0 and maximum is 40. For all subscales, minimum value is 0 and maximum is 10.
Changes in child's post-traumatic symptoms using the Revised Child Impact of Events Scale | Baseline, 12 months, 24 months
  Revised Child Impact of Events Scale (CRIES-8) is a 8-item child-friendly measure designed to screen children at risk for Post-Traumatic Stress Disorder (PTSD). the CRIES-8 has two sub-scales (Intrusion and Avoidance). Total scores range from 0 to 40, with higher scores indicated higher PTSD symptoms. A reduction in trauma symptoms would indicate improvement.
Change in child mental health using the Revised Children's Anxiety and Depression Scale (RCADS) | Baseline, 12 months, 24 months
  The Revised Children's Anxiety and Depression Scale (RCADS) is a self- and parent-reported measure that assesses a child's internalizing problems, specifically symptoms of anxiety and depression. Sub-scales assess for separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood (major depressive disorder). Results produce a total anxiety score and total internalizing score. Higher scores indicate worse outcomes and a greater severity of anxiety or depression. For the total scale, the maximum score is 141 and the minimum is 0. For the sub scales: Generalized Anxiety Disorder (0 to 15), Social Phobia (0 to 15), Separation Anxiety Disorder (0 to 15), Panic Disorder (0 to 15), Depression (0 to 24)

SECONDARY OUTCOMES:
Change in cognitive functioning using Cambridge Neuropsychological Test Automated Battery | Baseline, 12 months, 24 months
  Cambridge Neuropsychological Test Automated Battery (CANTAB) of computer-based non-linguistic tasks that provide understanding of brain functions (Attention, Cognitive Control-Response Inhibition, Impulsivity). Children complete Emotional Bias Task (min: 0, max: 15), Motor Screening Task (min: 0, max: 6000), Reaction Time (min: 0, max: 5100), Stockings of Cambridge (min: 0, max: 12), and Spatial Span (min: 2, max: 9). Higher scores indicate better outcomes.
Change in school attendance | Baseline, 12 months, 24 months
  School attendance is collected from teachers and school records. Minimum score is 0 and maximum is the number of days in the school year (varies).
Change in cognitive functioning using Wechsler Intelligence Scale for Children (Fifth Edition) | Baseline, 12 months, 24 months
  The Wechsler Intelligence Scale for Children (Fifth Edition) is an intelligence test designed to assess the cognitive abilities in children. Children complete Block Design task, which assesses ability to visualize and manipulate spatial forms. Maximum scaled score is 19. Minimum scaled score is 1. A higher score indicates a better outcome.
Change in grade average | Baseline, 12 months, 24 months
  Change in school grades is collected from school academic records (report cards). The minimum grade is 0 and the maximum is 5. Higher grades indicate better outcomes.
Change in school problem behavior | Baseline, 12 months, 24 months
  Problem behavior is measured as a composite score of a teacher-reported likert scale of the frequency of student behaviors in school: get into fights with other students, has conflicts with teachers, parents are called, sent to the principal's office, completes homework (reversed). The minimum is 0 and the maximum is 5. Higher score indicates worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Ismayilova, PhD, Principal Investigator — University of Chicago
Locations (2):
- Azerbaijan (2):
  - National Mental Health Centre under the Ministry of Health, Baku, Azerbaijan
  - Research and Education Center, Baku, Azerbaijan

IPD SHARING:
Plan to Share IPD: Yes
Datasets will be made available to any individual who makes a direct request to the PIs and indicates the data will be used for the purposes of research (per Code of Federal Regulation Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge.").
  Shared data will be free of identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects. Data will be shared in electronic format native to the software used by the Investigators; requestors are expected to handle converting electronic formats (though the Investigators will consider converting to tab-delimited text format if possible).
Supporting Information: Study Protocol
Time Frame: Once all of the data have been de-identified, cleaned, and validated, and main findings have been published, the Investigators expect to share data with the scientific community.
  Upon completion of the deliverable(s), the requestor will be instructed to destroy all copies of the data. If deliverables have not been produced yet, the agreement to share data will be revisited annually to decide to continue sharing or terminate the sharing agreement. If the Investigators determine that the sharing agreement should be terminated, the requestor will be instructed to destroy all copies of the data.
Access Criteria: The University of Chicago has a data sharing agreement that specifies the following conditions be met before data are shared:
  1. A formal research question is specified a priori;
  2. Names, affiliations, and roles of any other individuals who will access the shared data;
  3. The deliverable(s) (e.g., manuscript, conference presentation) are specified a priori;
  4. Proper credit and attribution-e.g., authorship, co-authorship, and order-for each deliverable are specified a priori;
  5. A statement indicating an understanding that the data can not be further shared with any additional individual(s) or parties without the PI's permission;
  6. Institutional Review Board (IRB) approval for use of the data (or documentation that IRB has determined the research is exempt);